CLINICAL TRIAL: NCT04089930
Title: Long-term Immunogenicity of a Live Attenuated Herpes Zoster Vaccine (Zostavax) in Patients With Systemic Lupus Erythematosus
Brief Title: Long-term Immunogenicity of a Live Herpes Zoster Vaccine in Systemic Lupus Erythematosus (SLE) Patients
Status: Completed | Type: Observational
Sponsor: Tuen Mun Hospital (Other Government)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Chiu Mok, Consultant, Tuen Mun Hospital
Other Study IDs: NTWC/REC/19088
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Lupus Erythematosus
Keywords: herpes zoster; vaccine; lupus
MeSH Terms: conditions — Herpes Zoster | interventions — Immunogenicity, Vaccine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccine: Those SLE patients who had been given herpes zoster vaccine in our original RCT
  Interventions: Diagnostic Test: Immunogenicity
- Placebo: Those SLE patients who had been given placebo vaccination in our original RCT
  Interventions: Diagnostic Test: Immunogenicity

INTERVENTIONS:
Diagnostic Test: Immunogenicity — anti-VZV IgG titer and cell-mediated immunity (VZV-stimulated T cell spots)

SUMMARY:
A recent randomized controlled trial (RCT) from our group has demonstrated safety and immune response (both humoral and cell-mediated) of the live-attenuated herpes zoster (HZ) vaccine (Zostavax) in stable systemic lupus erythematosus (SLE) patients with a previous history of HZ or varicella infection. An important research question is whether the immunogenicity of the HZ vaccine in SLE patients is long-lasting. There is no information in the literature regarding the long-term immunogenicity and safety of Zostavax in SLE patients. This prompts the current extension study which is planned to evaluate the long-term immunogenicity and efficacy of Zostavax in our original patient cohort.

DETAILED DESCRIPTION:
A recent RCT from our group has demonstrated safety and immune response (both humoral and cell-mediated) of the live-attenuated Zostavax in stable SLE patients with a previous history of HZ or varicella infection. An important research question is whether the immunogenicity of the HZ vaccine in SLE patients is long-lasting. There is no information in the literature regarding the long-term immunogenicity and safety of the HZ vaccine, Zostavax, in SLE patients.

Patients who had completed the original RCT and had been followed for 5 years since HZ vaccination or placebo injection were invited to participate in this extension study. Blood samples will be taken for a repeat assessment of the humoral and cell-mediated response to VZV at 5 years.

Outcomes of interest Primary outcome Difference between the two groups in the proportion of patients who have a persistent and 50% increase in IgG to VZV (humoral response to Zostavax) at 5 years compared to baseline Secondary outcomes

1. Difference between the two groups in the cell-mediated response to Zostavax at 4 years as compared to baseline
2. Vaccine efficacy - difference in the rate of clinical HZ reactivation between two groups of patients at 5 years
3. Vaccine safety - difference between the two groups in terms of SLE flares and new autoimmune phenomena at 5 years

ELIGIBILITY:
Inclusion Criteria:

1. SLE patients who fulfill ≥4 of the 1997 ACR or the 2012 SLICC/ACR criteria for SLE or healthy controls who had participated in the original RCT
2. Age ≥18 years
3. Having completed the original RCT of HZ vaccine vs placebo
4. Having been followed for 5 years since HZ vaccination or placebo injection
5. Willing to comply with all study procedures

Exclusion Criteria:

1. Patients who refuse to participate in this long-term extension study
2. Patients in the placebo group who have subsequently received HZ vaccination
3. Patients who cannot give a written consent (mentally incapable or illiterate)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: systemic lupus erythematosus (SLE) patients
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Humoral immune response to vaccine | 5 years after vaccination
  percentage and absolute change in anti-VZV IgG titer from baseline

SECONDARY OUTCOMES:
Cell-mediated immune response to vaccine | 5 years after vaccination
  percentage and absolute change in VZV-stimulated T cell response (T cell spots) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chi Chiu Mok, Principal Investigator — Tuen Mun Hospital
Locations (1):
- Department of Medicine, Tuen Mun Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No